CLINICAL TRIAL: NCT05318313
Title: Telerehabilitation Effectiveness for Individuals With Temporomandibular Disorders (TMD): A Non-Inferiority Study
Brief Title: Telerehabilitation for TMD
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: DENT-2022-30141
Record Dates: First submitted 2022-03-03; First posted 2022-04-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Disorder; TMJ Disc Displacement With Reduction; TMJ Disc Displacement Without Reduction; Masticatory Myofascial Pain; TMJ Arthralgia; TMD Headache
Keywords: Temporomandibular Disorders; TMD; telerehabilitation; telehealth; physical therapy; PT
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Telerehabilitation only: Participants choose to have all of their physical therapy provided virtually throughout the length of the study
  Interventions: Other: Telerehabilitation
- In-person only: Participants choose to have all of their physical therapy provided in-person throughout the length of the study
- Hybrid 1: The TR PT evaluation and follow-up visits in the initial 6 weeks will be performed via Zoom software and subsequent follow-up visits will switch to in person after 6 weeks
  Interventions: Other: Telerehabilitation
- Hybrid 2: The PT evaluation and follow-up visits in the initial 6 weeks will be performed in person and will switch to TR via Zoom software after 6 weeks
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The TR PT evaluation and follow-up visits will be performed via Zoom software
  Groups: Hybrid 1; Hybrid 2; Telerehabilitation only

SUMMARY:
This study will compare after physical therapy for Temporomandibular Disorders (TMD) performed either in-person or virtually using telerehabilitation. Comparing diagnostic reliability and quality-of-life outcomes in each group will determine (based on a 10% margin) whether delivering physical therapy via telerehabilitation is as good as standard in-person care for these individuals. Long term outcomes including patient satisfaction, cost-effectiveness analysis, and functional status will describe the feasibility of telerehabilitation as a management intervention for this population.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Referred to PT with ≥1 TMD subtype diagnosis
* PI has no previous knowledge of the participant's diagnosis
* Email access
* Possession of any device that can be positioned for hands-free TR visits (TR group only)
* Willingness and ability to comply with all study requirements and PT program
* Able to provide informed consent

Exclusion Criteria:

* Non-English speakers
* Permanent residence outside of the state of Minnesota (TR group only)
* Women in the last trimester of pregnancy
* Referred for post-surgical rehabilitation
* Severe chronic pain as identified by level 4 classification on the GCPS
* Current diagnosis or existence of the following conditions that can limit response to PT and participation in study activities:

  1. Neuropathic pain
  2. Fibromyalgia and/or generalized widespread pain on both sides of the body in ≥3 areas above and below the waist
  3. Rheumatoid arthritis or juvenile idiopathic arthritis
  4. Dystonia or other movement disorder
  5. Fractures and/or recent jaw or facial trauma
  6. Malignancies
  7. Current substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with at least one subtype of temporomandibular disorders by a TMD specialist at the University of Minnesota TMD, Orofacial Pain and Dental Sleep Medicine Clinic and referred for physical therapy at the same clinic.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Specialist diagnosis | Measured directly after the PT evaluation (Day 1)
  Diagnosis will be determined by putting clinical assessment results into the Brief Diagnostic Criteria for TMD (Brief DC/TMD) algorithm and getting one or more of 7 possible diagnoses: TMJ arthralgia (joint), Masticatory myofascial pain (muscle), TMJ disc displacement with reduction (joint), TMJ disc displacement without reduction (joint), TMJ arthritis (joint), TMD headache (muscle), other (neither). The diagnosis will be measured as one of four options: 1. joint; 2. muscle; 3. both; or 4. neither.
Diagnostic agreement | Measured directly after the PT evaluation (Day 1)
  Agreement data for each subject will be collected comparing two specialist diagnoses: dentist and physical therapist. Agreement about the diagnostic category will be recorded as a binary "yes/no" measure.
The Oral Health Impact Profile for TMD summary score | 6 weeks after intervention onset
  The OHIP-TMD is a condition-specific quality-of-life scale with 22 items and a 0-4 scoring option for each item. A higher score means lower quality-of life. The summary score after 6 weeks will be compared to the baseline summary score, and a score decrease ≥6.9 units will be considered evidence of therapy success. The proportion of therapy success in each group will be used for non-inferiority comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kahnert, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States